CLINICAL TRIAL: NCT00170027
Title: Safety and Efficacy of the CMI Magnetocardiograph Model 2409 for Diagnosing Coronary Heart Disease
Brief Title: Safety and Efficacy of MCG for Diagnosing Coronary Heart Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: CardioMag Imaging (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: 999-03
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2011-02-15 (Estimated); Status verified 2011-02

CONDITIONS: Myocardial Ischemia
MeSH Terms: conditions — Myocardial Ischemia

INTERVENTIONS:
Device: Magnetocardiograph

SUMMARY:
A magnetocardiograph (MCG) is a medical device capable of recording the magnetic fields that arise from the electrical activity of the heart. It was developed for the general purpose as a noninvasive, non-contact diagnostic tool of obstructive coronary artery disease (CAD), and especially of cardiac ischemia. The overall objective of the present study is to demonstrate the efficacy of this MCG device in the diagnosis of lack of oxygen to an area of the heart (as in an Heart attack) in patients presenting with chest pain.

DETAILED DESCRIPTION:
The CMI-2409 magnetocardiograph (MCG) is an FDA-approved medical device capable of noninvasive recording of magnetic fields arising from the electrical activity of the heart. This system was developed by CMI for the general purpose of noninvasive, non-contact diagnostics of obstructive coronary artery disease (CAD), and especially of cardiac ischemia. The overall objective of the present study is to demonstrate the efficacy of this MCG device and of the associated MCG method for the detection and diagnosis of ischemia in chest pain patients.

The primary objective is to demonstrate that the diagnostic accuracy of the MCG device and method is equivalent to or better than that of a standard 12-lead ECG for detecting the presence of ischemia in patients presenting with chest pain of unknown etiology. In this study the rest MCG data will be analyzed and compared to the results of a rest ECG.

ELIGIBILITY:
Subjects with chest pain syndrome or angina equivalent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2003-07; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Primary endpoint will be final clinical diagnosis of ischemia by the primary treating physician. This decision will be based upon evaluation of symptoms, clinical presentation, 12-lead ECG, cardiac enzymes (Troponin I or CKMB).

SECONDARY OUTCOMES:
1. Correlation of MCG with anatomic patency and TIMI flow on coronary angiography
2. Correlation of MCG with functional and laboratory tests

CONTACTS AND LOCATIONS:
Overall Officials: Peter A. Smars, M.D. EM, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Related Info — http://www.cardiomag.com/